CLINICAL TRIAL: NCT00546884
Title: Intervention to Improve Expression of End of Life Preferences for Homeless Persons
Acronym: SELPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0704S06282; NR/NINR NIH (Other: NINR); R01NR009815 (NIH)
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: End of Life; Advance Directives; Randomized controlled trial; End of life care; End of life advance care planning
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI (Placebo Comparator): The MI condition will expose participants to the provision of an advance directive and written instructions, roughly mimicking community standards and the requirements of the federal Patient Self Determination Act.
  Interventions: Behavioral: MI condition
- GI (Active Comparator): Subjects randomized to the GI group will be invited to meet individually with a health care professional specializing in EOL care
  Interventions: Behavioral: GI

INTERVENTIONS:
Behavioral: MI condition — Individuals randomized to this condition will be provided with written end of life educational materials an advance directive form, along with instructions to complete it.
  Arms: MI
Behavioral: GI — The GI condition will expose participants to education, guidance and counseling, and an advance directive tool.
  Arms: GI

SUMMARY:
The purpose of this study is to determine whether homeless individuals will complete a living will and whether guidance enhances rates of completion and to see whether filling out a living will has any impact on the care given at the end of life.

DETAILED DESCRIPTION:
Much research and effort have been directed towards improving end-of-life (EOL) care in the US. However, there is consensus that large gaps in knowledge remain regarding quality EOL care, most notably because previous research has focused on narrowly defined populations. There is little known about individuals who are from different ethnic, cultural, and socioeconomic backgrounds. There is some evidence that these individuals may desire and experience EOL care differently and may encounter barriers to obtaining this care. What is not known is what interventions are effective in these populations. This study addresses EOL care for homeless people, the most extreme examples of these overlooked populations. They have the greatest risk of death in the US, have unique perspectives of good EOL care, encounter significant barriers to care, and lack the resources and relationships assumed necessary for good EOL care. Despite this, there are no interventional studies determining whether EOL care can be improved in this population. Encouraging individuals to document preferences for EOL care through Advance Directives (ADs), has been central to efforts to improve EOL care. ADs, however, have been subject to conceptual and empirical criticism, particularly that they may not ultimately affect EOL care received. However, these shortcomings have been mainly demonstrated in specific and similar populations, and has not been addressed in underserved populations. There are reasons to believe that ADs and advance care planning have different utility and efficacy for homeless persons and are much desired in this population. This proposal builds upon four years of research, including an NIH/NINR-funded investigation, regarding EOL care, dying, and death. This research is some of the first work defining the concerns of homeless persons regarding EOL care and confirmed the relevance and potential of ADs in this population to impact EOL care positively. We seek to test an intervention to improve EOL care for homeless persons: 300 participants will be randomized into two arms, guided intervention (GI) and minimal intervention (MI). The GI condition will expose participants to education, guidance and counseling, and an AD tool, designated HELP (Appendix A), specifically designed for underserved and estranged populations to enhance autonomy and elicit preferences of EOL care. The MI condition will expose participants to the provision of HELP and instructions, mimicking community standards and the requirements of the federal PSDA.

Primary Aim 1: To determine whether homeless individuals will complete an AD and whether guidance enhances rates of completion. Hypothesis 1: We hypothesize that the MI will result in greater completion rate in this population than most others studied, and that the GI will result in a significantly greater rate than the MI - we anticipate a 20% completion rate in the MI condition and a 50% rate in the GI condition. Primary Aim 2: To determine whether completion of ADs by homeless individuals lead to their use during county hospital care encounters over 18 months after the intervention. Hypothesis 2: We hypothesize that when completed ADs exist, they will be used or documented as part of clinical care at least 70% of the time during county health care encounters.

It is important to test appropriate, reproducible interventions in underserved populations, and insights from this project will be significant in several ways: they will help address the EOL concerns of homeless persons, and provide the basis to address the needs of others who are disenfranchised from loved ones and/or receive fragmented, episodic care, such as the rural and urban poor, homebound persons, or undocumented persons.

ELIGIBILITY:
Inclusion Criteria:

* Homeless in the previous 6 months as defined by the federal McKinney Act
* At least 18 years old
* Speak English
* Able to give valid informed consent

Exclusion Criteria:

* Actively intoxicated
* Cognitive deficiencies using BLESSED tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Y Song, MD, MPH, MAT, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - VA Medical Center, Minneapolis, Minnesota

REFERENCES:
- [Derived] Song J, Ratner ER, Wall MM, Bartels DM, Ulvestad N, Petroskas D, West M, Weber-Main AM, Grengs L, Gelberg L. Effect of an End-of-Life Planning Intervention on the completion of advance directives in homeless persons: a randomized trial. Ann Intern Med. 2010 Jul 20;153(2):76-84. doi: 10.7326/0003-4819-153-2-201007200-00003. PMID 20643989

RESULTS

PARTICIPANT FLOW:
Groups:
- Minimal Intervention: The MI condition will expose participants to the provision of an advance directive and written instructions, roughly mimicking community standards and the requirements of the federal Patient Self Determination Act.
  MI condition: Individuals randomized to this condition will be provided with written end of life educational materials an advance directive form, along with instructions to complete it.
- Guided Intervention: Subjects randomized to the GI group will be invited to meet individually with a health care professional specializing in EOL care
  GI: The GI condition will expose participants to education, guidance and counseling, and an advance directive tool.
Period: Overall Study
Arm/Group | Minimal Intervention | Guided Intervention
Started | 145 | 117
Completed | 145 | 117
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimal Intervention | Guided Intervention | Total
Number analyzed (Participants) | 145 | 117 | 262
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 123 | 94 | 217
  >=65 years | 22 | 23 | 45
Age, Continuous [Mean (Full Range); unit: years] | 43.3 [19 to 68] | 43.1 [21 to 70] | 43.1 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 111 | 82 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 11 | 18
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 81 | 60 | 141
  White | 48 | 35 | 83
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 145 | 117 | 262

OUTCOME MEASURES:

1. Primary Outcome: Completion of Advance Directive
Description: Completing an advance directive for the individuals health care when they are not able to direct it themselves
Time Frame: 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intervention | Guided Intervention
Number analyzed (Participants) | 117 | 145
Participants | 15 | 55
Statistical Analysis 1: Comparison: Minimal Intervention vs Guided Intervention; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 4.16

ADVERSE EVENTS:
Arm/Group | Minimal Intervention | Guided Intervention
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/117
Other Adverse Events (participants affected / at risk) | 0/145 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No